CLINICAL TRIAL: NCT02102672
Title: Comprehensive Evaluation of Right Ventricular Function, Ventricular Remodeling and Micro RNA Profiling in Pulmonary Artery Hypertension: Effects of a Fatty Acid Oxidation Inhibitor
Brief Title: Trimetazidine in Pulmonary Artery Hypertension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-229
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo 1 pill bid, 3 months
- Trimetazidine (Experimental): Trimetazidine 35 mg bid for 3 months
  Interventions: Drug: Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine
  Other Names: Vastarel
  Arms: Trimetazidine

SUMMARY:
Pulmonary artery hypertension (PAH) is a chronic and progressive disease that affects 15 persons per million. Although current therapy has improve disease prognosis, PAH still has a poor survival, with a median survival of 2.8 years after diagnosis. In the last few years new key elements in PAH pathogenesis have been discovered, such as the role of metabolism in disease onset and progression. In fact, PAH pulmonary smooth muscle cells switch into a glycolytic phenotype which resembles the metabolism of cancer cells. The investigators hypothesis is that "fatty acid oxidation inhibition reverts the PAH adverse phenotype by restoring mitochondrial function and morphology, decreasing proliferation and restoring apoptosis susceptibility in pulmonary smooth muscle cells "

ELIGIBILITY:
Inclusion Criteria:

* PAH patients belonging to the following subgroups of the updated Dana Point Classification Group 1

  1. Idiopathic PAH
  2. Heritable PAH
  3. Drug or toxin-induced PAH
  4. PAH associated with connective tissue disease
  5. PAH associated to congenital heart disease with simple systemic-to-pulmonary shunt at least 1 year after surgical repair
  6. PAH associated to HIV infection
* Documented hemodynamic diagnosis of PAH by right ventricular catheterization performed any time prior to screening
* Signed informed consent

Exclusion Criteria:

* Patients belonging to the subgroups of the updated Dana Point Classification Group I not listed in the inclusion criteria
* Patients belonging to the groups 2-5 of the updated Dana Point Classification Group
* Moderate to severe chronic pulmonary obstructive disease
* Documented left ventricular dysfunction
* Severe renal impairment (Serum creatinine > 2.5 mg/dL)
* Patients who are receiving or have been receiving any investigational drugs within 1 month before the baseline visit
* Acute or chronic impairment (other than dyspnea) limiting the ability to comply with study requirements
* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements
* Life expectancy less than 12 months
* Females who are lactating or pregnant or those who plan to become pregnant during the study
* Known hypersensitivity to any of the excipients of the drug formulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in right ventricular (RV) function | 3 months
  Changes in RV function assessed by echo 3d (strain-strain rate)

SECONDARY OUTCOMES:
Changes in exercise capacity | 3 months
  Changes in exercise capacity assessed by 6 minute walk test
Changes in symptoms | 3 months
  Changes in Borg dyspnea index
Changes in biomarkers | 3 months
  Changes in B-type natriuretic peptide, galectin-3 and rho-kinase activity
Time to clinical worsening | 3 months
  Time to first PAH related medical event (ER evaluation, hospitalization or death)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo F Castro, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile